CLINICAL TRIAL: NCT04275973
Title: Evaluating Mobility Interventions in the Real World
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-0844; A196200 (Other: UW Madison); ENGR/MECHANICAL ENGR/MECH ENGR (Other: UW Madison); BA180043 (Other Grant/Funding Number: US Department of Defense); Protocol Version 9/21/2023 (Other: UW Madison)
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Lower Limb Amputation; Drop Foot
Keywords: Prostheses; Orthoses
MeSH Terms: conditions — Peroneal Neuropathies | interventions — Artificial Limbs; Orthotic Devices

STUDY DESIGN:
Intervention Model Description: Participants will perform testing inside the laboratory ("lab testing"), outside the laboratory ("field testing") on the campus of University of Wisconsin, Madison, and/or extended testing in a home and community environment ("take-home testing") to evaluate different aspects of device function.
  Outcomes will generally be compared using a repeated-measures design, in which each participant acts as his/her own control. This design is chosen to minimize the statistical problems caused by heterogeneity in the participant population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Prosthesis user with transtibial or transfemoral amputation (Experimental): Experiments will use standard commercially available prostheses for participants with lower-limb amputation. Specific prostheses will be determined at the time of the study, but they will include prostheses that are fully passive such as energy storage-and-return (ESR) feet, ESR feet with mobilized ankles such as passive hydraulic ankles (PHA), and ESR feet with microprocessor-controlled ankles (MPA).
  Interventions: Device: Lower limb prostheses
- Orthoses user with drop-foot (Experimental): This arm will consists of participants with drop-foot. A subset of the drop-foot population will be persons with Multiple Sclerosis and currently drop-foot.
  For participants in this arm, standard commercially-available orthoses or standard-of-care custom orthoses will be used, as well as standard commercially-available electrical stimulation neuro-orthoses.
  Interventions: Device: Orthoses for Drop-foot

INTERVENTIONS:
Device: Lower limb prostheses — Standard commercially available prostheses for participants with lower-limb amputation.
  Specific prostheses will be determined at the time of the study, but they will include prostheses that are fully passive such as energy storage-and-return (ESR, Agilix) feet and low-profile foot (LP, Pacifica LP), ESR feet with mobilized ankles such as passive hydraulic ankles (PHA, Kinterra), and ESR feet with microprocessor-controlled ankles (MPA, Kinnex).
  Other Names: Low-profile foot; Energy-storing foot; Hydraulic ankle; Microprocessor ankle
  Arms: Prosthesis user with transtibial or transfemoral amputation
Device: Orthoses for Drop-foot — Standard commercially-available orthoses or standard-of-care custom orthoses as well as standard commercially-available electrical stimulation neuro-orthoses.
  Sprystep for the caAFO, Bioness L300 Go for the FES
  Other Names: carbon fiber ankle foot orthosis (caAFO); functional electrical stimulation (FES)
  Arms: Orthoses user with drop-foot

SUMMARY:
This study is intended to test the comparative biomechanical benefits of different lower-limb prostheses and orthoses using data collected over extended periods of everyday life using wearable sensors. Investigators seek to improve physical health, functional activity level, independence, workforce participation, and mental health in participants with lower limb amputation and other lower-limb impairments. Investigators seek to study the similarities and differences in participants' movement using prostheses and orthoses with different technological features or designs. Study team also seek to develop technologies that enhance the methods for using wearable sensor technology to perform this type of study.

Participants with lower-limb amputation, participants who use lower limb orthoses, and participants with drop-foot (including a specific group with Multiple Sclerosis).

ELIGIBILITY:
Inclusion Criteria:

Target Populations:

* Participants with amputation must have used a prosthesis for more than 6 months, and wear it for at least 8 hours per day.
* Participants must be more than 6 months past their most recent surgery (if any).
* Participants must be free of musculoskeletal and cardiovascular conditions that would limit their ability to safely complete testing.
* Participants should consider themselves in good health; be able to wear their prostheses or orthoses all day long; be able to perform all of their activities of daily living (ADL) with their prostheses or orthoses as appropriate; have a comfortably fitting functional prosthesis (if applicable) that does not cause any skin problems; and have a stable residual limb (or impaired limb).
* Participants may use a narrow-base cane (single point, narrow tripod base, etc.) as an ambulatory aid but not a small-base quad cane or walker.
* Participants must be able to walk with their prostheses or orthoses for 30 minutes (total) and stand for 30 minutes (total), in individual bouts of at least 6 minutes, without becoming fatigued, feeling dizzy, having chest pain or shortness of breath, or experiencing claudication symptoms.
* Participants involved in running tests must be able to run for 30 minutes (total) in bouts of at least 6 minutes, without becoming fatigued, feeling dizzy, having chest pain, or experiencing claudication symptoms.
* Participants must have no known cognitive disability.
* Participants must be fluent in spoken and written English.
* Running portions of the study will be limited to participants who self-report regular engagement in recreational or competitive running.
* Participants in the branch that uses only their own prostheses must have at least a daily use prosthesis and a running-specific prosthesis; additional prostheses may also be included

Multiple Sclerosis group:

* For the specific subgroup targeting Multiple Sclerosis, participants must have a clinical diagnosis of Multiple Sclerosis and a clinician must determine they are experiencing foot drop.
* Participants must be able to comfortably wear and ambulate with both study devices with effective management of foot-drop, without significant discomfort
* Participants must be able to perform all of their activities of daily living (ADL) with only minimal use of ambulatory aids. Subjects may use a narrow-base cane (single point, narrow tripod base, etc.) as an ambulatory aid in any amount. Use of more comprehensive ambulatory aids (e.g. a small-base quad cane, wide-base quad cane or walker) must be limited to no more than 20% of their walking time when not at home. Participants who do use an assistive device occasionally should report a threshold for use of greater than 100 feet, i.e., they are unlikely to use their device unless they anticipate ambulating greater than this distance.

Exclusion Criteria:

Target Populations:

* Allergy to electrode gel, surgical tape and metals.
* Participants who currently use the Bioness L300 Go or similar neuro-orthoses or use a carbon fiber ankle-foot orthosis at the time of the study will be excluded to avoid biasing results for one device or the other. Participants with past experience not currently using these devices will be eligible.
* Participants enrolled in physical therapy or other rehabilitative care for treatment of gait, balance, or lower extremity strength or coordination at the time of the study will be excluded to avoid confounding effects from therapy and device-based management of their condition.
* For the orthotics study, participants with peripheral neuropathy impacting control of the tibialis anterior muscle via the peroneal nerve will be excluded.
* Participants under treatment for infectious diseases will be excluded from the study.
* Women who are pregnant or planning to become pregnant during the course of the study will be excluded.
* Symptomatic musculoskeletal conditions that prevent unaided walking, such as back pain or knee arthritis.
* Cardiovascular conditions that make moderate exercise unsafe, including (but not limited to) history of angina, peripheral vascular disease, congestive heart failure, history of myocardial infarction, and history of stroke. Potential participants will be excluded if they self-report that a physician has told them to avoid moderate exercise.
* History of chest pain, shortness of breath, or claudication symptoms during ambulation
* History of significant neuropathy with altered balance
* History of serious residual limb pain or phantom limb pain within the past six months.
* History of chronic skin breakdown.
* Inability to perform the tasks involved in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Adamczyk, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Healthy control participants were not consented or enrolled.
Groups:
- Prosthesis User With Transtibial or Transfemoral Amputation: Experiments will use standard commercially available prostheses for participants with lower-limb amputation. Specific prostheses will be determined at the time of the study, but they will include prostheses that are fully passive such as energy storage-and-return (ESR) feet, ESR feet with mobilized ankles such as passive hydraulic ankles (PHA), and ESR feet with microprocessor-controlled ankles (MPA).
  Lower limb prostheses: Standard commercially available prostheses for participants with lower-limb amputation.
  Specific prostheses will be determined at the time of the study, but they will include prostheses that are fully passive such as energy storage-and-return (ESR) feet, ESR feet with mobilized ankles such as passive hydraulic ankles (PHA), and ESR feet with microprocessor-controlled ankles (MPA).
- Orthoses User With Drop-foot: This arm will consists of participants with drop-foot. All of the drop-foot population were persons with Multiple Sclerosis.
  For participants in this arm, standard commercially-available orthoses or standard-of-care custom orthoses will be used, as well as standard commercially-available electrical stimulation neuro-orthoses.
  Orthoses for Drop-foot: Standard commercially-available orthoses or standard-of-care custom orthoses as well as standard commercially-available electrical stimulation neuro-orthoses.
Period: Overall Study
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation | Orthoses User With Drop-foot
Started | 8 | 12
Low Profile Foot | 5 | 0
Energy Storage and Return Foot | 5 | 0
Passive Hydraulic Ankle | 5 | 0
Microprocessor Hydraulic Ankle | 2 | 0
No Intervention | 0 | 11
Ankle Foot Orthosis (AFO) | 0 | 11
Functional Electrical Stimulation (FES) Device | 0 | 11
Completed | 6 | 11
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation | Orthoses User With Drop-foot | Total
Number analyzed (Participants) | 6 | 11 | 17
Age, Continuous [Mean (Full Range); unit: years] | 57 [44 to 67] | 43 [32 to 67] | 48 [32 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 6 | 11 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 11 | 17
Region of Enrollment [Number; unit: participants]
  United States | 6 | 11 | 17
Participants Diagnosed with Multiple Sclerosis (MS) [Count of Participants; unit: Participants] | 0 | 11 | 11

OUTCOME MEASURES:

1. Primary Outcome: Minimum Foot Clearance With Different Prostheses
Description: Minimum Foot Clearance with different prostheses, participants crossover to each of 4 different conditions at different study visits, data collected up to 12 weeks on study.
Time Frame: Weekly time points for Prosthetic interventions (baseline, 1, 2, 3, and 4 weeks), data collected anytime up to 12 weeks on study
Population: All participants did not complete tests with all prostheses.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation
Number analyzed (Participants) | 6
meters
  Low Profile Foot: number analyzed (Participants) | 5
  Low Profile Foot | 0.02117 (0.005247)
  Energy Storage and Return Foot: number analyzed (Participants) | 5
  Energy Storage and Return Foot | 0.01976 (0.007828)
  Passive Hydraulic Ankle: number analyzed (Participants) | 5
  Passive Hydraulic Ankle | 0.01932 (0.004138)
  Microprocessor Hydraulic Ankle: number analyzed (Participants) | 2
  Microprocessor Hydraulic Ankle | 0.03055 (0.001360)

2. Primary Outcome: Minimum Foot Clearance With Different Orthoses
Description: Minimum Foot Clearance with different orthoses, participants crossover to each of 3 different conditions at different study visits, data collected up to 20 days on study.
Time Frame: Baseline, 10 days, and 20 days for Orthotic interventions
Population: 1 participant could not be assessed for this measure
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Orthoses User With Drop-foot
Number analyzed (Participants) | 10
centimeters
  No Intervention | 0.56469 (0.662561)
  Ankle Foot Orthosis | 0.721081 (0.857378)
  Functional Electrical Stimulation Device | 0.81136 (1.105746)

3. Secondary Outcome: Behavioral Gait Function as Measured From Daily Stride Count
Description: Behavioral gait function will be measured by daily stride count (strides per sensor hour, Prosthetics only), participants crossed over to each of 4 different conditions at different study visits, data collected up to 12 weeks on study.
Time Frame: as for outcome 1
Population: All participants did not complete tests with all prostheses.
Measure: Mean (Standard Deviation); unit: strides per sensor hour
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation
Number analyzed (Participants) | 6
strides per sensor hour
  Low Profile Foot: number analyzed (Participants) | 5
  Low Profile Foot | 264.9 (177.0)
  Energy Storage and Return Foot: number analyzed (Participants) | 5
  Energy Storage and Return Foot | 245.7 (113.1)
  Passive Hydraulic Ankle: number analyzed (Participants) | 5
  Passive Hydraulic Ankle | 230.9 (117.8)
  Microprocessor Hydraulic Ankle: number analyzed (Participants) | 2
  Microprocessor Hydraulic Ankle | 269.3 (92.49)

4. Secondary Outcome: Behavioral Gait Function as Measured From Stride Speed During Walking Bouts of Different Durations
Description: Behavioral gait function will be measured by average stride speed, participants crossover to each of 4 different conditions at different study visits, data collected up to 12 weeks on study.
Time Frame: as for outcome 1
Population: Participants had varying ability to walk at different speeds.
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation
Number analyzed (Participants) | 6
meters per second
  less than 10 seconds | 0.4685 (0.049)
  10 to 30 seconds | 0.7155 (0.0936)
  30-60 seconds | 0.906 (0.1172)
  60-120 seconds: number analyzed (Participants) | 5
  60-120 seconds | 0.9652 (0.1562)
  greater than 120 seconds: number analyzed (Participants) | 4
  greater than 120 seconds | 1.0486 (0.1979)

5. Secondary Outcome: Prosthetic Limb Users Survey of Mobility Score
Description: The Prosthetic Limb Users Survey of Mobility (PLUS-M) is a 12 item questionnaire. It is a self-report instrument for measuring mobility of adults with lower limb amputation.
  PLUS-M instruments measure prosthetic users' mobility (i.e., the ability to move intentionally and independently from one place to another). PLUS-M questions assess respondents' perceived ability to carry out actions that require use of both lower limbs, ranging from household ambulation to outdoor recreational activities. The described activities relate to two primary forms of movement, locomotion (i.e., movement in a continuous, repeatable pattern) and/or postural transitions (i.e., movement from one position to another or one type of activity to another).
  PLUS-M instruments provide a T-score that averages 50 with a standard deviation of 10. A higher PLUS-M T-score corresponds to greater mobility.
Time Frame: up to 12 weeks
Population: All participants did not complete tests with all prostheses.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation
Number analyzed (Participants) | 6
T-score
  Low Profile Foot | 56.5 (7.665246245)
  Energy Storage and Return Foot | 53.78 (7.3123)
  Passive Hydraulic Ankle | 53.83 (7.898)
  Microprocessor Hydraulic Ankle: number analyzed (Participants) | 3
  Microprocessor Hydraulic Ankle | 47.4 (5.444)

6. Secondary Outcome: Change in Movement Quality as Determined by Stride Width: Prosthesis
Description: Change in movement quality will be determined by stride width, participants crossover to each of 4 different conditions at different study visits, data collected up to 12 weeks on study. Stride width is the absolute value of the lateral distance from a line that is fit to the foot placements of 3 strides previous and 3 strides after the current stride, to the foot placement location of the current stride.
Time Frame: as for outcome 1
Population: All participants did not complete tests with all prostheses.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation
Number analyzed (Participants) | 6
meters
  Low Profile Foot: number analyzed (Participants) | 5
  Low Profile Foot | 0.1328 (0.03138)
  Energy Storage and Return Foot: number analyzed (Participants) | 5
  Energy Storage and Return Foot | 0.1417 (0.05243)
  Passive Hydraulic Ankle: number analyzed (Participants) | 5
  Passive Hydraulic Ankle | 0.11526455 (0.02398894)
  Microprocessor Hydraulic Ankle: number analyzed (Participants) | 2
  Microprocessor Hydraulic Ankle | 0.1202 (0.04510)

7. Secondary Outcome: Change in Movement Quality as Determined by Stride Width: Orthoses
Description: Change in movement quality will be determined by stride width, participants crossover to different conditions at different study visits, data collected up to 20 days on study. Stride width is the absolute value of the lateral distance from a line that is fit to the foot placements of 3 strides previous and 3 strides after the current stride, to the foot placement location of the current stride.
Time Frame: Baseline, 10 days, and 20 days for Orthotic interventions
Population: Sensor did not work for one participant during the AFO condition.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Orthoses User With Drop-foot
Number analyzed (Participants) | 11
meters
  No Intervention | 0.045 (0.010)
  AFO: Sprystep: number analyzed (Participants) | 10
  AFO: Sprystep | 0.045 (0.010)
  FES: Bioness | 0.047 (0.014)
Statistical Analysis 1: Comparison: Orthoses User With Drop-foot; No Intervention vs AFO; Test type: Superiority; p = 0.649, t-test, 2 sided
Statistical Analysis 2: Comparison: Orthoses User With Drop-foot; No Intervention vs FES; Test type: Superiority; p = 0.513, t-test, 2 sided
Statistical Analysis 3: Comparison: Orthoses User With Drop-foot; AFO vs FES; Test type: Superiority; p = 0.617, t-test, 2 sided

8. Secondary Outcome: Change in Gait Performance as Determined by Average Speed
Description: Change in gait performance as determined by speed of the participant, participants crossover to each of 4 different conditions at different study visits, data collected up to 12 weeks on study.
Time Frame: as for outcome 1
Population: All participants did not complete tests with all prostheses.
Measure: Mean (Standard Deviation); unit: meter per second
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation
Number analyzed (Participants) | 6
meter per second
  Low Profile Foot: number analyzed (Participants) | 5
  Low Profile Foot | 0.8376 (0.1332)
  Energy Storage and Return Foot: number analyzed (Participants) | 5
  Energy Storage and Return Foot | 0.8553 (0.1149)
  Passive Hydraulic Ankle: number analyzed (Participants) | 5
  Passive Hydraulic Ankle | 0.8635 (0.1444)
  Microprocessor Hydraulic Ankle: number analyzed (Participants) | 2
  Microprocessor Hydraulic Ankle | 0.9521 (0.08561)

9. Secondary Outcome: Gait Performance as Determined by Stride Frequency at Identical Speed
Description: Gait performance as determined by stride frequency at identical speed (included strides with walking speeds between 0.75-1.25 meters per second). Participants crossover to each of 4 different conditions at different study visits, data collected up to 12 weeks on study.
Time Frame: as for outcome 1
Population: All participants did not complete tests with all prostheses.
Measure: Mean (Standard Deviation); unit: strides per minute
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation
Number analyzed (Participants) | 6
strides per minute
  Low Profile Foot: number analyzed (Participants) | 5
  Low Profile Foot | 67.47 (3.237)
  Energy Storage and Return Foot: number analyzed (Participants) | 5
  Energy Storage and Return Foot | 68.22 (5.835)
  Passive Hydraulic Ankle: number analyzed (Participants) | 5
  Passive Hydraulic Ankle | 67.46 (4.130)
  Microprocessor Hydraulic Ankle: number analyzed (Participants) | 2
  Microprocessor Hydraulic Ankle | 60.37 (5.448)

10. Secondary Outcome: Change in Gait Performance as Determined by Ground Reaction Forces
Description: Ground reaction force is force applied by the body to the ground. Peak forces and shape of the force vs. time trajectory are commonly used to assess gait quality. Forces closer to "normal" are usually considered better, but this goal does not apply in participants with amputation.
Time Frame: Baseline, 10 days, and 20 days for Orthotic interventions, weekly time points for Prosthetic interventions (baseline, 1, 2, 3, and 4 weeks), data collected anytime up to 12 weeks on study
Population: No data was collected because the force and torque sensor could not be fit into the leg.
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation | Orthoses User With Drop-foot
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Gait Performance as Determined by Socket Torques
Description: Socket torque (also termed "socket moment") is the amount of twisting or bending torque applied to the prosthetic socket. Peak socket torque and cumulative socket torque are measures commonly used to assess gait quality in persons with lower limb amputation.
Time Frame: as for outcome 10
Population: No data collected because the force and torque sensor could not be fit into the leg.
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation | Orthoses User With Drop-foot
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Functional Gait Assessment Score
Description: The Functional Gait Assessment Score will be measured for the sub-population of participants with Multiple Sclerosis (MS). The total score ranges from 0-30 with higher scores indicating increased impairment in gait. Participants crossover to each of three conditions at different study visits.
Time Frame: Baseline, 10 days, and 20 days for Orthotic interventions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Orthoses User With Drop-foot
Number analyzed (Participants) | 11
score on a scale
  No Intervention | 16.09 (5.230)
  Ankle Foot Orthosis | 17.27 (6.566)
  Functional Electrical Stimulation Device | 18.45 (5.298)

13. Secondary Outcome: Change in 6 Minute Walking Test Distance
Description: The sub-population of participants with MS will undergo a 6 minute walking test for distance. Each participant will crossover to three conditions over three study visits: No intervention, the carbon fiber ankle foot orthosis (cfAFO), and a functional electrical stimulation (FES) device). Reported here are the difference from No intervention for the cfAFO and FES orthoses, a positive number shows an increase in distance walked due to the intervention.
Time Frame: Baseline, 10 days, and 20 days study visits to test conditions for Orthotic interventions
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Orthoses User With Drop-foot
Number analyzed (Participants) | 11
meters
  No Intervention | 394.94 (123.83)
  AFO: Sprystep | 426.73 (117.87)
  FES: Bioness | 419.09 (127.16)

14. Secondary Outcome: Stride Length at Identical Walking Speed
Description: Walking speeds from 0.75 to 1.25 meters per second were analyzed, participants crossover to each of 4 different conditions at different study visits, data collected up to 12 weeks on study.
Time Frame: as for outcome 1
Population: All participants did not complete tests with all prostheses.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation
Number analyzed (Participants) | 6
meters
  Low Profile Foot: number analyzed (Participants) | 5
  Low Profile Foot | 1.196 (0.1434)
  Energy Storage and Return Foot: number analyzed (Participants) | 5
  Energy Storage and Return Foot | 1.198 (0.09409)
  Passive Hydraulic Ankle: number analyzed (Participants) | 5
  Passive Hydraulic Ankle | 1.200 (0.1564)
  Microprocessor Hydraulic Ankle: number analyzed (Participants) | 2
  Microprocessor Hydraulic Ankle | 1.302 (0.1194)

ADVERSE EVENTS:
Time Frame: participants were on study up to 12 weeks
Arm/Group | Prosthesis User With Transtibial or Transfemoral Amputation | Orthoses User With Drop-foot
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/11
Other Adverse Events (participants affected / at risk) | 0/6 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT04275973/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT04275973/ICF_000.pdf